CLINICAL TRIAL: NCT06800092
Title: Sildenafil to Prevent and Reduce Cancer Related Cognitive Impairment
Acronym: SPARC
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-0247
Record Dates: First submitted 2025-01-15; First posted 2025-01-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Fatigue; Brain Fog
MeSH Terms: conditions — Neoplasms; Fatigue; Mental Fatigue | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care Treatment (No Intervention): standard of care treatment
- Standard of Care Treatment and Sildenafil (Experimental): Sildenafil, 50mg, daily for duration of the standard of care treatment
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Sildenafil, 50mg, daily
  Other Names: Viagra
  Arms: Standard of Care Treatment and Sildenafil

SUMMARY:
This study is examining the effects of standard of care cancer treatment as well as a medication called Sildenafil, on the cancer associated fatigue, cognition and the gut microbiome.

DETAILED DESCRIPTION:
Cancer related cognitive impairment (CRCI) severely impacts neurocognitive function and is characterized by deficits in memory, learning, processing speed, and executive function. This cognitive impairment commonly referred to as "brain fog" or "chemo-brain," often co-occurs with central and peripheral fatigue. Symptoms typically begin acutely with the initiation of therapy, and persist chronically throughout prolonged treatment. Despite advancements in cytotoxic chemotherapies, CRCI plagues 75% of breast cancer patients during treatment, and development of new therapeutic options have been hampered by an incomplete understanding of the underlying mechanisms that cause CRCI. Although the etiology is not clear, CRCI is known to be associated with oxidative stress, increased inflammation, and disruption to the blood-brain barrier (BBB). Importantly, the endothelial cells of the BBB protect the central nervous system (CNS) from harmful and inflammatory bloodborne factors. Similarly, endothelial and epithelial barriers in the gut prevent microbial invasion and resulting regional and systemic inflammatory signaling. Thus, gut and brain barriers regulate exposure of the CNS to inflammatory factors and represent an important source of communication in the gut-brain axis. Research suggests that cytotoxic chemotherapeutic agents compromise both brain and gut endothelial and epithelial barrier integrity, leading to extravasation of toxins and immune cells into the CNS, causing neuroinflammation and CRCI. This study proposes that sildenafil, a phosphodiesterase-5 (PDE-5) inhibitor, will preserve barrier integrity during chemotherapy by downregulating oxidative and nitrosative stress that leads to endothelial dysfunction via multiple pathways. Thus, the goal of this project is to interrogate how chemotherapy-induced brain and gut barrier dysfunction mediate CRCI, neurotoxicity, and neuro- and systemic inflammation. Outcomes will be measured at baseline and throughout standard of care treatment, specifically after neoadjuvant chemotherapy, surgery, radiation treatment, chemotherapy treatment and after 24 weeks of endocrine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 30 - 50 years
* Self-reported menses occurrence within past 12 months
* Diagnosis of ER+/HER2- breast cancer
* Willing and able to comply with study procedures
* Willing and able to provide consent

Exclusion Criteria:

* Untreated thyroid disorder
* Untreated diabetes
* BMI >30
* Current treatment with metformin
* Diagnosed neuromuscular disease
* Diagnosed neurovascular disease
* Prior history of cognitive impairment
* Prior history of chemotherapy treatment
* HIV, Hepatitis B or Hepatitis C
* Systolic blood pressure <90 or >170, diastolic blood pressure <50 or >110 after repeated evaluation with proper cuff. This range is the acceptable range stated in the prescribing information for sildenafil (>90/50 and <170/110)
* Use of alpha blockers in the past 2 weeks
* Use of PDE5 inhibitors in the past 2 weeks
* Use of nitrates
* Subjects with MRI incompatible devices
* Subjects with severe claustrophobia
* Any medical condition that, in the opinion of the investigator, would place the subject at increased risk for participation

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female only
Enrollment: 30 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue and Cognition as measured by the Fatigue and Altered Cognition Scale at baseline | Baseline
  The Fatigue and Altered Cognition Scale (FACS) is a joint project from University of Texas Medical Branch and Texas A&M University. The FACS is a 20 question assessment designed to access perceived fatigue and cognition. There are 2 subscales used to calculate a total score. The subscales are: Fatigue and Altered Cognition. The total score is calculated by adding the subscales together. The range of the total score is 0-100, with a higher score indicating more fatigue and altered cognition.
Fatigue and Cognition as measured by the Fatigue and Altered Cognition Scale after neoadjuvant chemotherapy treatment | through neoadjuvant chemotherapy treatment completion, average of 20 weeks from baseline
  The Fatigue and Altered Cognition Scale (FACS) is a joint project from University of Texas Medical Branch and Texas A&M University. The FACS is a 20 question assessment designed to access perceived fatigue and cognition. There are 2 subscales used to calculate a total score. The subscales are: Fatigue and Altered Cognition. The total score is calculated by adding the subscales together. The range of the total score is 0-100, with a higher score indicating more fatigue and altered cognition.
Fatigue and Cognition as measured by the Fatigue and Altered Cognition Scale after surgery | through completion of surgery, average of 24 weeks from baseline
  The Fatigue and Altered Cognition Scale (FACS) is a joint project from University of Texas Medical Branch and Texas A&M University. The FACS is a 20 question assessment designed to access perceived fatigue and cognition. There are 2 subscales used to calculate a total score. The subscales are: Fatigue and Altered Cognition. The total score is calculated by adding the subscales together. The range of the total score is 0-100, with a higher score indicating more fatigue and altered cognition.
Fatigue and Cognition as measured by the Fatigue and Altered Cognition Scale after radiation treatment | through radiation treatment completion, average of 30 weeks from baseline
  The Fatigue and Altered Cognition Scale (FACS) is a joint project from University of Texas Medical Branch and Texas A&M University. The FACS is a 20 question assessment designed to access perceived fatigue and cognition. There are 2 subscales used to calculate a total score. The subscales are: Fatigue and Altered Cognition. The total score is calculated by adding the subscales together. The range of the total score is 0-100, with a higher score indicating more fatigue and altered cognition.
Fatigue and Cognition as measured by the Fatigue and Altered Cognition Scale after chemotherapy treatment | through chemotherapy treatment completion, average of 50 weeks from baseline
  The Fatigue and Altered Cognition Scale (FACS) is a joint project from University of Texas Medical Branch and Texas A&M University. The FACS is a 20 question assessment designed to access perceived fatigue and cognition. There are 2 subscales used to calculate a total score. The subscales are: Fatigue and Altered Cognition. The total score is calculated by adding the subscales together. The range of the total score is 0-100, with a higher score indicating more fatigue and altered cognition.
Fatigue and Cognition as measured by the Fatigue and Altered Cognition Scale after 24 weeks of endocrine treatment | through 24 weeks of endocrine treatment, average of 74 weeks from baseline
  The Fatigue and Altered Cognition Scale (FACS) is a joint project from University of Texas Medical Branch and Texas A&M University. The FACS is a 20 question assessment designed to access perceived fatigue and cognition. There are 2 subscales used to calculate a total score. The subscales are: Fatigue and Altered Cognition. The total score is calculated by adding the subscales together. The range of the total score is 0-100, with a higher score indicating more fatigue and altered cognition.
Perceived Cognition measured by the Functional Assessment of Cancer Therapy - Cognitive (FACT-Cog) at baseline | baseline
  The FACT-Cog is a self-administered measure of perceived cognitive impairment for patients undergoing cancer therapy. The FACT-Cog (version 3) contains 37 items which quantify 4 subscale domains using a 5 point Likert-type scale including: perceived cognitive impairments, impact of perceived cognitive impairments on quality of life, comments from others and perceived cognitive abilities. Perceived cognitive impairments subscale will be reported (range: 0-72, with a higher score indicating better quality of life).
Perceived Cognition measured by the Functional Assessment of Cancer Therapy - Cognitive (FACT-Cog) after neoadjuvant chemotherapy treatment | through neoadjuvant chemotherapy treatment completion, average of 20 weeks from baseline
  The FACT-Cog is a self-administered measure of perceived cognitive impairment for patients undergoing cancer therapy. The FACT-Cog (version 3) contains 37 items which quantify 4 subscale domains using a 5 point Likert-type scale including: perceived cognitive impairments, impact of perceived cognitive impairments on quality of life, comments from others and perceived cognitive abilities. Perceived cognitive impairments subscale will be reported (range: 0-72, with a higher score indicating better quality of life).
Perceived Cognition measured by the Functional Assessment of Cancer Therapy - Cognitive (FACT-Cog) after surgery | through completion of surgery, average of 24 weeks from baseline
  The FACT-Cog is a self-administered measure of perceived cognitive impairment for patients undergoing cancer therapy. The FACT-Cog (version 3) contains 37 items which quantify 4 subscale domains using a 5 point Likert-type scale including: perceived cognitive impairments, impact of perceived cognitive impairments on quality of life, comments from others and perceived cognitive abilities. Perceived cognitive impairments subscale will be reported (range: 0-72, with a higher score indicating better quality of life).
Perceived Cognition measured by the Functional Assessment of Cancer Therapy - Cognitive (FACT-Cog) after radiation treatment | through radiation treatment completion, average of 30 weeks from baseline
  The FACT-Cog is a self-administered measure of perceived cognitive impairment for patients undergoing cancer therapy. The FACT-Cog (version 3) contains 37 items which quantify 4 subscale domains using a 5 point Likert-type scale including: perceived cognitive impairments, impact of perceived cognitive impairments on quality of life, comments from others and perceived cognitive abilities. Perceived cognitive impairments subscale will be reported (range: 0-72, with a higher score indicating better quality of life).
Perceived Cognition measured by the Functional Assessment of Cancer Therapy - Cognitive (FACT-Cog) after chemotherapy treatment | through chemotherapy treatment completion, average of 50 weeks from baseline
  The FACT-Cog is a self-administered measure of perceived cognitive impairment for patients undergoing cancer therapy. The FACT-Cog (version 3) contains 37 items which quantify 4 subscale domains using a 5 point Likert-type scale including: perceived cognitive impairments, impact of perceived cognitive impairments on quality of life, comments from others and perceived cognitive abilities. Perceived cognitive impairments subscale will be reported (range: 0-72, with a higher score indicating better quality of life).
Perceived Cognition measured by the Functional Assessment of Cancer Therapy - Cognitive (FACT-Cog) after 24 weeks of endocrine therapy treatment | through 24 weeks of endocrine treatment, average of 74 weeks from baseline
  The FACT-Cog is a self-administered measure of perceived cognitive impairment for patients undergoing cancer therapy. The FACT-Cog (version 3) contains 37 items which quantify 4 subscale domains using a 5 point Likert-type scale including: perceived cognitive impairments, impact of perceived cognitive impairments on quality of life, comments from others and perceived cognitive abilities. Perceived cognitive impairments subscale will be reported (range: 0-72, with a higher score indicating better quality of life).
Perceptual Fatigue as measured by the MD Anderson Brief Fatigue Inventory (BFI) at baseline | baseline
  Perceptual fatigue will be assessed using the Brief Fatigue Inventory (BFI), a 9-item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life). The scores from all 9 questions can be average to calculate a Global Fatigue Score, with a range from 0 to 10, with a higher score indicating more fatigue.
Perceptual Fatigue as measured by the MD Anderson Brief Fatigue Inventory (BFI) after neoadjuvant chemotherapy treatment | through neoadjuvant chemotherapy treatment completion, average of 20 weeks from baseline
  Perceptual fatigue will be assessed using the Brief Fatigue Inventory (BFI), a 9-item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life). The scores from all 9 questions can be average to calculate a Global Fatigue Score, with a range from 0 to 10, with a higher score indicating more fatigue.
Perceptual Fatigue as measured by the MD Anderson Brief Fatigue Inventory (BFI) after surgery | through completion of surgery, average of 24 weeks from baseline
  Perceptual fatigue will be assessed using the Brief Fatigue Inventory (BFI), a 9-item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life). The scores from all 9 questions can be average to calculate a Global Fatigue Score, with a range from 0 to 10, with a higher score indicating more fatigue.
Perceptual Fatigue as measured by the MD Anderson Brief Fatigue Inventory (BFI) after radiation treatment | through radiation treatment completion, average of 30 weeks from baseline
  Perceptual fatigue will be assessed using the Brief Fatigue Inventory (BFI), a 9-item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life). The scores from all 9 questions can be average to calculate a Global Fatigue Score, with a range from 0 to 10, with a higher score indicating more fatigue.
Perceptual Fatigue as measured by the MD Anderson Brief Fatigue Inventory (BFI) after chemotherapy treatment | through chemotherapy treatment completion, average of 50 weeks from baseline
  Perceptual fatigue will be assessed using the Brief Fatigue Inventory (BFI), a 9-item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life). The scores from all 9 questions can be average to calculate a Global Fatigue Score, with a range from 0 to 10, with a higher score indicating more fatigue.
Perceptual Fatigue as measured by the MD Anderson Brief Fatigue Inventory (BFI) after 24 weeks of endocrine treatment | through 24 weeks of endocrine treatment, average of 74 weeks from baseline
  Perceptual fatigue will be assessed using the Brief Fatigue Inventory (BFI), a 9-item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life). The scores from all 9 questions can be average to calculate a Global Fatigue Score, with a range from 0 to 10, with a higher score indicating more fatigue.

SECONDARY OUTCOMES:
Quantify absolute abundance of gut microbiome using using metagenomic analysis at baseline | baseline
  Metagenomic analysis using a custom PCR array will be performed on stool samples to identify associated changes in microbiome absolute abundance at the genus and species level.
Quantify absolute abundance of gut microbiome using metagenomic analysis after neoadjuvant chemotherapy treatment | through neoadjuvant chemotherapy treatment completion, average of 20 weeks from baseline
  Metagenomic analysis using a custom PCR array will be performed on stool samples to identify associated changes in microbiome absolute abundance at the genus and species level.
Quantify absolute abundance of gut microbiome using metagenomic analysis after surgery | through completion of surgery, average of 24 weeks from baseline
  Metagenomic analysis using a custom PCR array will be performed on stool samples to identify associated changes in microbiome absolute abundance at the genus and species level.
Quantify absolute abundance of gut microbiome using metagenomic analysis after radiation treatment | through radiation treatment completion, average of 30 weeks from baseline
  Metagenomic analysis using a custom PCR array will be performed on stool samples to identify associated changes in microbiome absolute abundance at the genus and species level.
Quantify absolute abundance of gut microbiome using metagenomic analysis after chemotherapy treatment | through chemotherapy treatment completion, average of 50 weeks from baseline
  Metagenomic analysis using a custom PCR array will be performed on stool samples to identify associated changes in microbiome absolute abundance at the genus and species level.
Quantify absolute abundance of gut microbiome using metagenomic analysis after 24 weeks of endocrine treatment | through 24 weeks of endocrine treatment, average of 74 weeks from baseline
  Metagenomic analysis using a custom PCR array will be performed on stool samples to identify associated changes in microbiome absolute abundance at the genus and species level.
Fold change in relative abundance of gut microbiome using using metatranscriptomic analysis from baseline to after neoadjuvant chemotherapy treatment | through neoadjuvant chemotherapy treatment completion, average of 20 weeks from baseline
  Metatranscriptomic analysis using a RNA seq will be performed on stool samples to identify associated fold changes in which genes are turned on and off
Fold change in relative abundance of gut microbiome using using metatranscriptomic analysis from baseline to after surgery | through completion of surgery, average of 24 weeks from baseline
  Metatranscriptomic analysis using a RNA seq will be performed on stool samples to identify associated fold changes in which genes are turned on and off
Fold change in relative abundance of gut microbiome using using metatranscriptomic analysis from baseline to after radiation treatment | through radiation treatment completion, average of 30 weeks from baseline
  Metatranscriptomic analysis using a RNA seq will be performed on stool samples to identify associated fold changes in which genes are turned on and off
Fold change in relative abundance of gut microbiome using using metatranscriptomic analysis from baseline to after chemotherapy treatment | through chemotherapy treatment completion, average of 50 weeks from baseline
  Metatranscriptomic analysis using a RNA seq will be performed on stool samples to identify associated fold changes in which genes are turned on and off
Fold change in relative abundance of gut microbiome using using metatranscriptomic analysis from baseline to after 24 weeks of endocrine treatment | through 24 weeks of endocrine treatment, average of 74 weeks from baseline
  Metatranscriptomic analysis using a RNA seq will be performed on stool samples to identify associated fold changes in which genes are turned on and off

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Sheffield-Moore, PhD, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States